CLINICAL TRIAL: NCT01655680
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Parallel-Group, Phase 2 Study of the Safety and Efficacy of ABT-126 in the Treatment of Cognitive Deficits in Schizophrenia (CDS) in Nonsmokers
Brief Title: A Study to Evaluate ABT-126 for the Treatment of Cognitive Deficits in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-855; 2012-000418-13 (EudraCT Number)
Record Dates: First submitted 2012-05-25; First posted 2012-08-02 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ABT-126 Low Dose (Experimental): ABT-126 Low Dose
  Interventions: Drug: ABT-126
- ABT-126 Middle Dose (Experimental): ABT-126 Middle Dose
  Interventions: Drug: ABT-126
- ABT-126 High Dose (Experimental): ABT-126 High Dose
  Interventions: Drug: ABT-126
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-126 — ABT-126 Middle Dose
  Arms: ABT-126 Middle Dose
Drug: ABT-126 — ABT-126 Low Dose
  Arms: ABT-126 Low Dose
Drug: ABT-126 — ABT-126 High Dose
  Arms: ABT-126 High Dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a safety and efficacy study evaluating a experimental treatment for cognitive deficits in adults with schizophrenia.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to evaluate the safety and efficacy of ABT-126 in treating cognitive deficits in subjects with a diagnosis of schizophrenia. Eligible subjects will take study drug as an add-on treatment to their ongoing antipsychotic treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Has a current Diagnostic and Statistical Manual of Mental Disorders-, 4th Edition, Text Revision (DSM-IV-TR) diagnosis of schizophrenia confirmed by the Mini-International Neuropsychiatric Interview (M.I.N.I.).
* Is clinically stable while receiving a regimen of one or two allowable antipsychotic medications: lack of hospitalizations in 4 months prior to initial screening visit; taking the same antipsychotic medication(s) for at least 8 weeks prior to baseline visit; core positive symptoms of Positive and Negative Syndrome Scale (PANSS) no worse than moderate in severity throughout screening period of at least 4 weeks.
* Has been diagnosed with or treated for schizophrenia for at least 2 years prior to initial screening visit.
* Has had continuity in psychiatric care (e.g., mental health system, clinic or physician) for at least 6 months prior to initial screening visit.
* Has an identified contact person (e.g., family member, social worker, case worker, or nurse) that can provide support to the subject to ensure compliance with protocol requirements.

Exclusion Criteria:

* In the Investigator's judgment, has a current or past diagnosis of schizoaffective disorder, bipolar disorder, manic episode, dementia, post traumatic stress disorder, or obsessive-compulsive disorder, or the subject has a current major depressive episode.
* Has a positive urine drug screen for cocaine, phencyclidine (PCP), opiates (unless duly prescribed), benzodiazepines (unless duly prescribed), marijuana, or amphetamines during the Screening Period.
* Has a current or past history of seizures, with the exception of a single febrile seizure occurring prior to 6 years of age.
* Has a clinically significant abnormal electrocardiogram (ECG) at Screening Visit 1 as determined by the Investigator.
* Has any risk factors for Torsades de Pointes (TdP)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Cognition: MCCB (MATRICS Consensus Cognitive Battery) | Change from baseline to week 24
  Rater based interview

SECONDARY OUTCOMES:
Functioning: UPSA-2 (University of California San Diego Performance-based Skills Assessment-2) | Measurements from screening period up through week 24
  Rater based interview
Symptom Severity: PANSS (Positive and Negative Symptom Scale) | Measurements from screening period up through week 24
  Rater based interview
Symptom Severity: NSA-16 (16-item version of the Negative Symptom Assessment Scale) | Measurements from screening period up through week 24
  Rater based interview

CONTACTS AND LOCATIONS:
Overall Officials: George Haig, PharmD, Study Director — AbbVie
Locations (61):
- United States (34):
  - Site Reference ID/Investigator# 75139, Anaheim, California
  - Site Reference ID/Investigator# 74894, Bellflower, California
  - Site Reference ID/Investigator# 74434, Chino, California
  - Site Reference ID/Investigator# 76593, Costa Mesa, California
  - Site Reference ID/Investigator# 73213, Escondido, California
  - Site Reference ID/Investigator# 72698, Garden Grove, California
  - Site Reference ID/Investigator# 75057, La Habra, California
  - Site Reference ID/Investigator# 72693, National City, California
  - Site Reference ID/Investigator# 77655, Norwalk, California
  - Site Reference ID/Investigator# 74895, Oakland, California
  - Site Reference ID/Investigator# 73977, Oceanside, California
  - Site Reference ID/Investigator# 73214, Orange, California
  - Site Reference ID/Investigator# 74453, Pico Rivera, California
  - Site Reference ID/Investigator# 74898, Riverside, California
  - Site Reference ID/Investigator# 98016, San Bernardino, California
  - Site Reference ID/Investigator# 86973, San Diego, California
  - Site Reference ID/Investigator# 75140, San Diego, California
  - Site Reference ID/Investigator# 73974, San Gabriel, California
  - Site Reference ID/Investigator# 74433, Santa Ana, California
  - Site Reference ID/Investigator# 72695, Torrance, California
  - Site Reference ID/Investigator# 75136, New Haven, Connecticut
  - Site Reference ID/Investigator# 75653, Atlanta, Georgia
  - Site Reference ID/Investigator# 74893, Marietta, Georgia
  - Site Reference ID/Investigator# 72697, Chicago, Illinois
  - Site Reference ID/Investigator# 76533, Hoffman Estates, Illinois
  - Site Reference ID/Investigator# 75056, Wichita, Kansas
  - Site Reference ID/Investigator# 72694, Cedarhurst, New York
  - Site Reference ID/Investigator# 75137, Rochester, New York
  - Site Reference ID/Investigator# 75053, Staten Island, New York
  - Site Reference ID/Investigator# 75413, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 74553, Dallas, Texas
  - Site Reference ID/Investigator# 72696, DeSoto, Texas
  - Site Reference ID/Investigator# 75055, Houston, Texas
  - Site Reference ID/Investigator# 74896, Houston, Texas
- Russia (20):
  - Site Reference ID/Investigator# 94476, Chita
  - Site Reference ID/Investigator# 94528, Kazan'
  - Site Reference ID/Investigator# 79517, Lipetsk
  - Site Reference ID/Investigator# 81934, Moscow
  - Site Reference ID/Investigator# 81935, Moscow
  - Site Reference ID/Investigator# 79516, Moscow
  - Site Reference ID/Investigator# 83116, Novosibirsk
  - Site Reference ID/Investigator# 80673, Saint Petersburg
  - Site Reference ID/Investigator# 85093, Saint Petersburg
  - Site Reference ID/Investigator# 97135, Saint Petersburg
  - Site Reference ID/Investigator# 97137, Saint Petersburg
  - Site Reference ID/Investigator# 83115, Saint Petersburg
  - Site Reference ID/Investigator# 97136, Saint Petersburg
  - Site Reference ID/Investigator# 84733, Saint Petersburg
  - Site Reference ID/Investigator# 81933, Saratov
  - Site Reference ID/Investigator# 79514, Saratov
  - Site Reference ID/Investigator# 79520, Stavropol
  - Site Reference ID/Investigator# 83117, Yaroslavl
  - Site Reference ID/Investigator# 97138, Yekaterinburg
  - Site Reference ID/Investigator# 79515, Yekaterinburg
- United Kingdom (7):
  - Site Reference ID/Investigator# 81938, Brentford
  - Site Reference ID/Investigator# 81940, Edinburgh
  - Site Reference ID/Investigator# 81939, London
  - Site Reference ID/Investigator# 92813, London
  - Site Reference ID/Investigator# 81937, Newcastle upon Tyne
  - Site Reference ID/Investigator# 81943, Oxford
  - Site Reference ID/Investigator# 82238, Preston

REFERENCES:
- [Result] Haig G, Wang D, Othman AA, Zhao J. The alpha7 Nicotinic Agonist ABT-126 in the Treatment of Cognitive Impairment Associated with Schizophrenia in Nonsmokers: Results from a Randomized Controlled Phase 2b Study. Neuropsychopharmacology. 2016 Nov;41(12):2893-2902. doi: 10.1038/npp.2016.101. Epub 2016 Jun 20. PMID 27319970
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500
- [Derived] Bain EE, Shafner L, Walling DP, Othman AA, Chuang-Stein C, Hinkle J, Hanina A. Use of a Novel Artificial Intelligence Platform on Mobile Devices to Assess Dosing Compliance in a Phase 2 Clinical Trial in Subjects With Schizophrenia. JMIR Mhealth Uhealth. 2017 Feb 21;5(2):e18. doi: 10.2196/mhealth.7030. PMID 28223265